CLINICAL TRIAL: NCT03371589
Title: Intratympanic Stereoidal Injections for Facial Nerve Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0057-17
Record Dates: First submitted 2017-05-29; First posted 2017-12-13 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients who cannot receive the oral treatment due to a prior condition e.g. diabetes, high blood pressure, pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- no P.O corticosteroids (Experimental): Steroids injection
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Solution for otic injection

SUMMARY:
Bell's palsy is defined as a facial nerve palsy without any other known cause. The common practice for this disease consists of the use of oral steroids. Such treatment can cause harm to people who have disabilities or prior conditions such as pregnancies, diabetes, obesity and/or high blood pressure. While the use of intratympanic injection for sudden sensory hearing loss is well rehearsed in many practices, similar management of facial nerve palsy due to Bell's phenomenon is rare and a few researches have been conducted regarding the subject. In this research we suggest intratympanic injections for these patients as a treatment for Bell's palsy.

DETAILED DESCRIPTION:
Bell's palsy is defined as a facial nerve paralysis without any other known diagnosis or cause .Its' estimated occurrence is in 20 to 30 people per 100,000 people per year. The occurence is greater in patients older than 65 years old and lower in children younger than 13 years old. There are many estimated etiologies for Bell's palsy, such as failure of the vasa nervosa, viral infections, ischemic neuropathies and auto immune reactions. Of those, viral hypothesis is the most widely accepted.

The prognosis for recovery for most patients is 80% to 90%. One series showed that only 17 out of 1505 patients demonstrated moderate to severe sequela and none had complete facial nerve paralysis. The common practice for the management of Bell's palsy consists of oral steroids with or without the antiviral medications. A recent study made by the Department of Otorhinolaryngology and Head and Neck surgery in Korea indicated that Intratympanic injections could replace the use of oral steroids . Another recent study by Jong job lee et al. has shown that Intratympanic injections have prolonged uptake in rats, in comparison to Intraperitoneal injections.

ELIGIBILITY:
Inclusion Criteria:

Adult patients 18 years old or more, diagnosed with Bell's palsy who cannot receive oral steroid treatment for their condition, due to to pregnancy, diabetes, high blood pressure etc.

Exclusion Criteria:

* Children under the age of 18.
* Patients who can receive oral steroid treatment for their condition.
* Patients with internal ear problems. * Patients who already recieved treatmetn for their condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
House brackman scale | change in score 1 month, 3 months and 6 months after end of treatment
  grade 1-6

SECONDARY OUTCOMES:
Nottingham scale for facial palsy | change in score 1 month, 3 months and 6 months after end of treatment
  ratio (distance between point in the face in cm)

CONTACTS AND LOCATIONS:
Overall Officials: Muhamad Taha, MD, Principal Investigator — Hillel Yaffe MC

IPD SHARING:
Plan to Share IPD: Undecided